CLINICAL TRIAL: NCT07320326
Title: A Multi-center, Ambispective, Non-interventional, Observational, Registry Study of the Effectiveness of Elranatamab in Patients With Triple-class Exposed Relapsed/Refractory Multiple Myeloma in Routine Clinical Practice in China(ASPIRE: A Registry Study Of Chinese Patients With TCE-RRMM Treated By Elranatamab)
Brief Title: ASPIRE: A Registry Study Of Chinese Patients With TCE-RRMM Treated By Elranatamab
Acronym: ASPIRE
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jin Lu, MD, Dr, Peking University People's Hospital
Other Study IDs: ID#98552787
Record Dates: First submitted 2025-12-09; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: TCE-RRMM
Keywords: TCE-RRMM; Elranatamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Elranatamab treatment cohort: In the retrospective period, Each patient will be followed up until two years after the first dose of Elranatamab treatment, death, or withdrawal of consent, whichever occurs first. Information collection will be performed every month for the first 6 months after the first dose of Elranatamab treatment and then every 3 months for the following 18 months.
  The prospective period will include a Screening Period and a Treatment Period. Screening Period assessments will be performed within 7 days prior to treatment. During the Treatment Period, each patient will be followed up until two years after the first dose of Elranatamab treatment, death, or withdrawal of consent, whichever occurs first.
  Interventions: Drug: Elranatamab

INTERVENTIONS:
Drug: Elranatamab — In the retrospective period, Each patient will be followed up until two years after the first dose of Elranatamab treatment, death, or withdrawal of consent, whichever occurs first. Information collection will be performed every month for the first 6 months after the first dose of Elranatamab treatment and then every 3 months for the following 18 months. The prospective period will include a Screening Period and a Treatment Period. Screening Period assessments will be performed within 7 days prior to treatment. During the Treatment Period, each patient will be followed up until two years after the first dose of Elranatamab treatment, death, or withdrawal of consent, whichever occurs first.

SUMMARY:
This registry study will provide valuable evidence to assess and validate its effectiveness in the Chinese MM population, refine clinical application strategies, and support the optimization of BCMA BsAbs use in MM treatment in China.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignancy characterized by the clonal proliferation of terminally differentiated plasma cells within the bone marrow. It is the second most common hematological malignancy, accounting for 10-15% of all hematological cancers. Over the past three to four decades, the incidence of MM has been increasing globally. Similar trends are observed in China, where the incidence of MM has also been rising. According to the GLOBOCAN database, in 2022, there were an estimated 30,300 new cases of MM and 18,662 deaths. The 5-year prevalence rate was approximately 6.0 per 100,000 people in China.

Remarkable progress in MM has been achieved in the past two decades. Proteasome inhibitors (PIs), immunomodulatory drugs (IMiDs), and anti-CD38 monoclonal antibodies (mAbs) are the cornerstone of MM therapeutics. After the incorporation of three class novel agents the clinical outcomes of patients with MM have improved significantly, however, MM remains incurable, as most patients eventually experience relapse/progression. Relapse and progression remain the primary causes of mortality in MM patients.

As relapses are common in MM, and patients often receive various drug combinations throughout the course of their disease, providing optimal therapy for patients already exposed to PIs, IMiDs, and anti-CD38 mAbs s (namely triple-class exposed [TCE]) and/or refractory to these drugs (triple-class refractory [TCR]) presents a significant therapeutic challenge. The LocoMMotion and MAMMOTH studies have highlighted the dismal outcomes of patients with TCE/TCR MM, with response rates of approximately 30% and a complete response (CR) or better (<1%). Furthermore, the progression-free survival (PFS) and overall survival (OS) for this patient subset are limited, with a median PFS of no longer than 6 months and median OS of less than 1 year. As a result, there is an urgent and increasing unmet need for novel therapies with new targets, mechanisms of action, and treatment strategies to extend the duration and durability of clinical responses, thereby improving survival outcomes for TCE/TCR MM patients.

BMCA is a member of the tumor necrosis factor (TNF) receptor superfamily and plays a crucial role in the survival of long-lived bone marrow plasma cells (PCs). Additionally, the overexpression of serum BCMA correlates with disease progression and shorter PFS and OS in patients with MM, making BCMA an ideal therapeutic target. Recently, immunotherapies targeting BCMA have shown promise in the treatment of relapsed or refractory multiple myeloma (RRMM). The chimeric antigen receptor (CAR) T cell and bispecific antibodies (BsABs) targeting BCMA are emerging as a new standard of care in TCE-RRMM population. To date, two bispecific antibodies targeting CD3 on T cells and BCMA on myeloma cells have been approved globally for the treatment of TCE-RRMM patients.

Elranatamab, a humanized BCMA-CD3 BsAB was granted accelerated approval by the FDA in August 2023 for the treatment of patients with TCE-RRMM, based on the results of the MagnetisMM-3 (NCT04649359) study. In the MagnetisMM-3 study (Cohort A), elranatamab led to an ORR of 61%, with a median PFS of 17.2 months in TCE-RRMM patients who had received a median of 5 prior lines of therapy. The median duration of response (DOR) was not reached, with a median follow-up of 33.9 months. Elranatamab was approved by the National Medical Products Administration (NMPA) in March 2025 in China. However, real-world data on its use in the Chinese population is currently lacking, and physicians have limited experience administering it outside of clinical trials.

Therefore, collecting real-world data on the effectiveness of Elranatamab in Chinese TCE-RRMM patients after its commercially available in China is crucial.

ELIGIBILITY:
Inclusion Criteria:

Participants with TCE-RRMM who have received or are planning to start Elranatamab treatment according to the local Health Authority approved product label (routine-care).

Patients must meet the following criteria to be eligible for inclusion in the study:

In the retrospective part:

1. Male or female patients above 18 years old
2. Patients diagnosed with RRMM(IMWG)
3. Prior lines of therapy must include a proteasome inhibitor, an immunomodulatory drug and anti-CD38 monoclonal antibody in any order during the course of treatment
4. Patients received at least 1 treatment dose of Elranatamab treatment after commercial launch in China and according to the approved product label (routine-care) in China (consistent with the approved label in China)*
5. Patients understand and voluntarily sign an ICF .

In the prospective part:

1. Male or female patients above 18 years old
2. Patients diagnosed with RRMM (IMWG)
3. Prior lines of therapy must include a proteasome inhibitor, an immunomodulatory drug and anti-CD38 monoclonal antibody in any order during the course of treatment
4. Patients treated with elranatamab as monotherapy or a part of combination therapy and according to the approved product label (routine-care) in China (consistent with the approved label in China)*
5. Patient understand and voluntarily sign an ICF. *Note: If patients received Elranatamab treatment at a Hong Kong site,the treatment must consist the indications approved in Hong Kong.

Exclusion Criteria:

Patients meeting the following criteria will not be included in the study:

In the retrospective part:

1. Patients with documented diagnosis of other cancers prior to the diagnosis of MM
2. Patients enrolled in interventional clinical trials of any drug for MM treatment
3. Patients with incomplete medical records or missing clinical laboratory data that preclude effectiveness evaluation.
4. Patients who, in the opinion of the investigator, have other factors that make them unsuitable for study participation.

In the prospective part:

1. Patients with documented diagnosis of other cancers prior to the diagnosis of MM
2. Patients with contraindication listed in the package insert of elranatamab
3. Patients enrolled in interventional clinical trials of Elranatamab or any other drug for MM treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with TCE-RRMM who have received or are planning to start Elranatamab treatment according to the local Health Authority approved product label (routine-care).
  Patients must meet the Inclusion Criteria and the Exclusion Criteria to be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-07-18 (Estimated); Study Completion 2028-09-18 (Estimated)

PRIMARY OUTCOMES:
ORR | At the time from the date of first dose until the first documentation of PD, death or start of new anticancer therapy, whichever occurs first , assessed up to 27 months.
  Overall Response Rate (ORR):(including PR, VGPR, CR, and sCR)

SECONDARY OUTCOMES:
PFS | As the time from the date of first dose until PD per IMWG criteria or death due to any cause, whichever occurs first, assessed up to 27 months.
  Progression-freesurvival
OS | As the time from the date of first dose until death due to any cause, assessed up to 27 months.
  Overall survival
DOR | As the time from the first documentation of objective response that is subsequently confirmed, until PD per IMWG criteria, or death due to any cause, whichever occurs first, assessed up to 27 months.
  Duration of response
MRD negativity rate | The proportion of participants in the analysis population with negative MRD per IMWG criteria by BMA at any time after first dose, assessed up to 27 months.
  Minimal Residual Disease negativity rate
TTR | For participants with an objective response per IMWG criteria, as the time from the date of first dose to the first documentation of objective response that is subsequently confirmed, assessed up to 27 months.
  Time to response
PRO: EORTC QLQ-C30、EORTC QLQ-MY20 and EQ-5D-5L will be used in this study | From the screening visit to the last follow up visit, assessed up to 27 months.
  To evaluate the patient-reported outcomes of Elranatamab-treated TCE-RRMM patients in China using the following patient-reported outcome (PRO) instruments:
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Version 3.0 (EORTC QLQ-C30) European Organization for Research and Treatment of Cancer Multiple Myeloma Questionnaire (EORTC QLQ-MY20) The EuroQol 5-Dimension 5-level (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Unplanned

REFERENCES:
- [Result] Kumar et al, 2016
- [Result] Cocks K, Cohen D, Wisloff F, Sezer O, Lee S, Hippe E, Gimsing P, Turesson I, Hajek R, Smith A, Graham L, Phillips A, Stead M, Velikova G, Brown J; EORTC Quality of Life Group. An international field study of the reliability and validity of a disease-specific questionnaire module (the QLQ-MY20) in assessing the quality of life of patients with multiple myeloma. Eur J Cancer. 2007 Jul;43(11):1670-8. doi: 10.1016/j.ejca.2007.04.022. Epub 2007 Jun 15. PMID 17574838
- [Result] Osoba D, Aaronson N, Zee B, Sprangers M, te Velde A. Modification of the EORTC QLQ-C30 (version 2.0) based on content validity and reliability testing in large samples of patients with cancer. The Study Group on Quality of Life of the EORTC and the Symptom Control and Quality of Life Committees of the NCI of Canada Clinical Trials Group. Qual Life Res. 1997 Mar;6(2):103-8. doi: 10.1023/a:1026429831234. PMID 9161109
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Result] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Result] Tomasson MH, Iida S, Niesvizky R, Mohty M, Bahlis NJ, Martinez-Lopez J, Koehne G, Rodriguez-Otero P, Miles Prince H, Viqueira A, Leip E, Conte U, Sullivan ST, Lesokhin AM. Long-term survival and safety of elranatamab in patients with relapsed or refractory multiple myeloma: Update from the MagnetisMM-3 study. Hemasphere. 2024 Jul 24;8(7):e136. doi: 10.1002/hem3.136. eCollection 2024 Jul. No abstract available. PMID 39055646
- [Result] Lesokhin AM, Tomasson MH, Arnulf B, Bahlis NJ, Miles Prince H, Niesvizky R, Rodriotaguez-Otero P, Martinez-Lopez J, Koehne G, Touzeau C, Jethava Y, Quach H, Depaus J, Yokoyama H, Gabayan AE, Stevens DA, Nooka AK, Manier S, Raje N, Iida S, Raab MS, Searle E, Leip E, Sullivan ST, Conte U, Elmeliegy M, Czibere A, Viqueira A, Mohty M. Elranatamab in relapsed or refractory multiple myeloma: phase 2 MagnetisMM-3 trial results. Nat Med. 2023 Sep;29(9):2259-2267. doi: 10.1038/s41591-023-02528-9. Epub 2023 Aug 15. PMID 37582952
- [Result] Tacchetti P, Barbato S, Mancuso K, Zamagni E, Cavo M. Bispecific Antibodies for the Management of Relapsed/Refractory Multiple Myeloma. Cancers (Basel). 2024 Jun 26;16(13):2337. doi: 10.3390/cancers16132337. PMID 39001399
- [Result] Holstein SA, Grant SJ, Wildes TM. Chimeric Antigen Receptor T-Cell and Bispecific Antibody Therapy in Multiple Myeloma: Moving Into the Future. J Clin Oncol. 2023 Sep 20;41(27):4416-4429. doi: 10.1200/JCO.23.00512. Epub 2023 Jul 20. PMID 37471687
- [Result] Sanchez L, Dardac A, Madduri D, Richard S, Richter J. B-cell maturation antigen (BCMA) in multiple myeloma: the new frontier of targeted therapies. Ther Adv Hematol. 2021 Jan 30;12:2040620721989585. doi: 10.1177/2040620721989585. eCollection 2021. PMID 33796236
- [Result] Cornelis R, Chang HD, Radbruch A. Keeping up with the stress of antibody production: BAFF and APRIL maintain memory plasma cells. Curr Opin Immunol. 2021 Aug;71:97-102. doi: 10.1016/j.coi.2021.06.012. Epub 2021 Jul 22. PMID 34303157
- [Result] Gandhi UH, Cornell RF, Lakshman A, Gahvari ZJ, McGehee E, Jagosky MH, Gupta R, Varnado W, Fiala MA, Chhabra S, Malek E, Mansour J, Paul B, Barnstead A, Kodali S, Neppalli A, Liedtke M, Narayana S, Godby KN, Kang Y, Kansagra A, Umyarova E, Scott EC, Hari P, Vij R, Usmani SZ, Callander NS, Kumar SK, Costa LJ. Outcomes of patients with multiple myeloma refractory to CD38-targeted monoclonal antibody therapy. Leukemia. 2019 Sep;33(9):2266-2275. doi: 10.1038/s41375-019-0435-7. Epub 2019 Mar 11. PMID 30858549
- [Result] Mateos MV, Weisel K, De Stefano V, Goldschmidt H, Delforge M, Mohty M, Cavo M, Vij R, Lindsey-Hill J, Dytfeld D, Angelucci E, Perrot A, Benjamin R, van de Donk NWCJ, Ocio EM, Scheid C, Gay F, Roeloffzen W, Rodriguez-Otero P, Broijl A, Potamianou A, Sakabedoyan C, Semerjian M, Keim S, Strulev V, Schecter JM, Vogel M, Wapenaar R, Nesheiwat T, San-Miguel J, Sonneveld P, Einsele H, Moreau P. LocoMMotion: a prospective, non-interventional, multinational study of real-life current standards of care in patients with relapsed and/or refractory multiple myeloma. Leukemia. 2022 May;36(5):1371-1376. doi: 10.1038/s41375-022-01531-2. Epub 2022 Mar 24. PMID 35332278
- [Result] Puertas B, Fernandez-Sanchez A, Alejo E, Rey-Bua B, Martin-Lopez AA, Perez-Lopez E, Lopez-Parra M, Lopez-Corral L, Gutierrez-Gutierrez NC, Garcia-Sanz R, Puig N, Gonzalez-Calle V, Mateos MV. A research center's experience of T-cell-redirecting therapies in triple-class refractory multiple myeloma. Blood Adv. 2024 Jul 9;8(13):3478-3487. doi: 10.1182/bloodadvances.2024012773. PMID 38717869
- [Result] Ahmed A, Killeen RB. Relapsed and Refractory Multiple Myeloma. 2023 Jun 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK592405/ PMID 37276320
- [Result] Bhatt P, Kloock C, Comenzo R. Relapsed/Refractory Multiple Myeloma: A Review of Available Therapies and Clinical Scenarios Encountered in Myeloma Relapse. Curr Oncol. 2023 Feb 15;30(2):2322-2347. doi: 10.3390/curroncol30020179. PMID 36826140
- [Result] Hu Q, Xiang B. Recent Advances in the Treatment of Multiple Myeloma in the Era of New Drug Development. Asp Biomed Clin Case Rep. 2024; 7(3):294-303
- [Result] Dou X, Duan G, Zhong Y, Liu Y, Peng N, Wen L, Qi J, Zhou M, Zhang X, Lu J. The burden of multiple myeloma in China: Trends from 1990 to 2021 and forecasts for 2050. Cancer Lett. 2025 Jan 2;611:217440. doi: 10.1016/j.canlet.2025.217440. Online ahead of print. PMID 39755360
- [Result] Malard F, Neri P, Bahlis NJ, Terpos E, Moukalled N, Hungria VTM, Manier S, Mohty M. Multiple myeloma. Nat Rev Dis Primers. 2024 Jun 27;10(1):45. doi: 10.1038/s41572-024-00529-7. PMID 38937492
- See also: World Health Organization. Globocan 2022: Multiple Myeloma. Available from: https://gco.iarc.who.int/media/globocan/factsheets/populations/160-china-fact-sheet.pdf [[Last accessed: March 2025]] — https://gco.iarc.who.int/media/globocan/factsheets/populations/160-china-fact-sheet.pdf